CLINICAL TRIAL: NCT04459494
Title: Evaluation of Dental Implant Treatment With and Without Flap for Clinical, Radiographic and Patient Comfort
Brief Title: In the Treatment of Implants With Different Methods; Early Bone Loss and Patient Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Erkan SARI, Research Assistant Dentist, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20164753772
Record Dates: First submitted 2020-07-02; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Dental Implants
Keywords: Dental Implants; marginal bone loss; flapless implant surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Patients undergoing dental implant treatment without flap removal (Test Group)
  Interventions: Procedure: Flapless implant surgery.
- Control group (Active Comparator): Patients who will receive dental implants by removing conventional full thickness flaps (Control group)
  Interventions: Procedure: Conventional implant surgery.

INTERVENTIONS:
Procedure: Flapless implant surgery. — Local anesthesia will be applied to the patients in the test group, and then the implant socket will be prepared without removing the flap and a dental implant will be placed.
  Bite-wing film will be taken to control the implants in the same session after surgery, and patients will be given VAS (visual analog scale) to perform their assessment of pain on the 3rd day and 7th day. Patients will be given an appointment again after 3 months of treatment. In this session, implants will be evaluated with bite-wing film.
  Arms: Test group
Procedure: Conventional implant surgery. — Local anesthesia will be applied to the patients in the control group, and then the implant socket will be prepared after reflecting the flap and a dental implant will be placed.
  Patients in the control group will receive a full thickness flap elevation and an implant socket will be prepared afterwards the implant will be placed and then the flap will be closed with 4-0 silk suture.
  Bite-wing film will be taken from both groups to control the implants in the same session after surgery, and patients will be given VAS (visual analog scale) to perform their assessment of pain on the 3rd day and 7th day. Patients will be given an appointment again after 3 months of treatment. In this session, implants will be evaluated with bite-wing film.
  Arms: Control group

SUMMARY:
The aim of this clinical study is to compare two different approaches during dental implant applications. One group of patients in the study received flapless approach which is performed without surgical reflection of soft tissues (gums) during implant surgery. In the control group of the study, patients received conventional flap approach in which flap reflections performed on soft tissues (gums) of the patients.

After the surgery patients were monitored for marginal bone loss around implants and discomfort after the surgery for 3 months. And received data statistically analyzed to compare the different surgical procedures.

DETAILED DESCRIPTION:
Filling the Case Report Form for each registered patient and signed by the responsible investigator or an authorized representative of the study staff. This also applies to records for patients who could not complete the study (even if a case report form was prepared, even during screening prior to randomization). If a patient withdraws from the study, the reason for this is recorded in the Case report form. If a patient withdraws from the study because of a limiting adverse event, all necessary efforts will be made to clearly document the result.

All forms must be filled with a typewriter or an indelible ink pen and must be readable. Errors can be crossed out, but errors cannot be deleted; the correction is entered and the change is initialed and dated by the investigator or his authorized representative. The researcher should ensure the accuracy, completeness and legibility of the data reported to the sponsor in the case report forms and all required reports and that it was processed on time.

The researcher is responsible for the accuracy of the data transferred on the forms and will sign these forms in the sense of showing their compatibility with the recorded data.

As a result of the power analysis made with G * Power3.1 (Franz Faul, UniversitätKiel, Germany) software program, it has been determined that the sampling number consisting of 20 people with 0.8 effect size and α = 0.05 significance level generates more than 80% power. it was deemed appropriate to include a total of 24 people in the study. Karim M. Ahmed A, Salah Abd Elfatah B, Mohamed Abd El-Mageed Katamish's ''Crestal bone loss of standard implant versus platform switch implant design using minimal invasive technique'' article is used as a reference for marginal bone loss data calculation.

Patients with sufficient amount of bone were included in the study after bone sounding and x rays were evaluated after local anesthesia before surgery. By an unbiased researcher, the patients were recruited to the groups using the envelope method; control group (with flap raised) or test group (without flap raised) were assigned.

A total of 24 patients complying with these criteria were included in the study and a total of 37 implants were applied to the patients.

Implant applications of the patients in the control group were performed by lifting the flap. The implants of the patients included in the test group were applied without lifting the flap.

For each implant in the study marginal bone loss were evaluated; Digital bite-wing x-rays taken with a standard technique were used.Bite-wing x-rays taken were standardized with bite blocks on the film holder prepared individually for each patient. From each implant site; two x-rays were taken first immediately after implant surgery and the second three months later, just before the uncovering session of the implants. Digital bite-wing x-rays were transferred to RadiAnt Dicom Viewer program and measurements were made on them. Implant diameter values which is known in the images are accepted as reference.The diameter in the image was measured and a coefficient was obtained by dividing the real diameter to measurement on image. In the images, the distance between the most coronal point of the implant neck and the point where the implant bone contact first occurred was measured. This distance was divided by the coefficient obtained and its actual values are obtained in mm.The difference between these distances at two time points were recorded in patient forms as marginal bone loss. In statistical analysis, comparisons between groups were made.

All the individuals included in the study came to the control appointments on the 3rd and 7th days after implant surgery, and the sutures were also taken on the 7th day. All patients were asked to fill the Turkish translation of Oral Health Impact Profile (OHIP-14) forms three times: preoperatively, postoperative day 3, and postoperative day 7. Visual Analog Scale (VAS) forms were asked to be marked by the patients on the 3rd and 7th days after the operation. VAS forms were prepared as a horizontal line with one side being the lowest score and the other side with highest score. VAS forms were prepared to be in 0-100 mm and the point marked by the patient was measured in cm. In VAS forms, patients were asked to mark according to their post-operative pain status.

Statistical analysis of the data in this study was done with Statistical Package for the Social Sciences (SPSS) 20 (International Business Machines Corporation Somers, New York, USA) package program.In the evaluation of the data, besides descriptive statistical methods (mean, standard deviation), T test was used for comparisons between groups. ANOVA test was used for multiple group comparisons. Statistical significance level was determined as p <0.05 .

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy (The determination of healthy volunteers will be based on the patient's statements in the anamnesis received. Additional examinations will not be performed.)
* Not smoking,
* Does not have a medication that he constantly uses,
* who have not used antibiotics, anti-inflammatory and systemic corticosteroid drugs in the last 6 months,
* Patients who are not in pregnancy, lactation, menstruation or menopause,
* Patients with at least 1 tooth deficiency,
* Patients who accepted the research and signed the informed volunteer consent form

Exclusion Criteria:

* Regularly using a systemic medication,
* During pregnancy, lactation, menstruation or menopause,
* Have any oral or systemic diseases,
* Receiving antibiotic, anti-inflammatory or systemic corticosteroid drug treatment in the last 6 months,
* Patients with no teeth deficiency

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Early marginal bone loss around implant neck. | Immediately after implant placement - 3 months after surgery.
  Bite wing x-rays taken with parallel technique for both groups were evaluated and recorded between the baseline and the 3rd month around the implant neck.

SECONDARY OUTCOMES:
Visual analog scale -Patient discomfort after surgery. | Immediately after implant surgery - 3 days after surgery - 7 days after surgery .
  Patients were given questionnaire for assessment of discomfort after surgery.
The Turkish translation of Oral Health Impact Profile (OHIP-14) forms - Patient discomfort after surgery. | Immediately after implant surgery - 3 days after surgery - 7 days after surgery .
  Patients were given questionnaire for assessment of discomfort after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Şükrü ENHOŞ, Study Director — Izmir Katip Celebi University Faculty of Dentistry
Locations (1):
- Izmir Katip Celebi University Faculty of Dentistry, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
patient privacy

REFERENCES:
- [Background] Sclar AG. Guidelines for flapless surgery. J Oral Maxillofac Surg. 2007 Jul;65(7 Suppl 1):20-32. doi: 10.1016/j.joms.2007.03.017. PMID 17586346
- [Background] Costich ER, Ramfjord SP. Healing after partial denudation of the alveolar process. J Periodontol. 1968 May;39(3):127-34. doi: 10.1902/jop.1968.39.3.127. No abstract available. PMID 5240004
- [Background] Staffileno H. Significant differences and advantages between the full thickness and split thickness flaps. J Periodontol. 1974 Jun;45(6):421-5. doi: 10.1902/jop.1974.45.6.421. No abstract available. PMID 4525958
- [Background] Rocci A, Martignoni M, Gottlow J. Immediate loading in the maxilla using flapless surgery, implants placed in predetermined positions, and prefabricated provisional restorations: a retrospective 3-year clinical study. Clin Implant Dent Relat Res. 2003;5 Suppl 1:29-36. doi: 10.1111/j.1708-8208.2003.tb00013.x. PMID 12691648
- [Background] Becker W, Goldstein M, Becker BE, Sennerby L. Minimally invasive flapless implant surgery: a prospective multicenter study. Clin Implant Dent Relat Res. 2005;7 Suppl 1:S21-7. doi: 10.1111/j.1708-8208.2005.tb00071.x. PMID 16137084
- [Background] Rao W, Benzi R. Single mandibular first molar implants with flapless guided surgery and immediate function: preliminary clinical and radiographic results of a prospective study. J Prosthet Dent. 2007 Jun;97(6 Suppl):S3-S14. doi: 10.1016/S0022-3913(07)60003-1. PMID 17618931
- [Background] Becker W, Goldstein M, Becker BE, Sennerby L, Kois D, Hujoel P. Minimally invasive flapless implant placement: follow-up results from a multicenter study. J Periodontol. 2009 Feb;80(2):347-52. doi: 10.1902/jop.2009.080286. PMID 19186977
- [Background] Arisan V, Karabuda CZ, Ozdemir T. Implant surgery using bone- and mucosa-supported stereolithographic guides in totally edentulous jaws: surgical and post-operative outcomes of computer-aided vs. standard techniques. Clin Oral Implants Res. 2010 Sep;21(9):980-8. doi: 10.1111/j.1600-0501.2010.01957.x. Epub 2010 May 24. PMID 20497439